CLINICAL TRIAL: NCT03133572
Title: Neonatal Supraglottic Airway Trial: A Single-centre, Open-label, Randomized Clinical Trial to Evaluate the Efficacy of I-gel® Supraglottic Airway Used in Neonatal Resuscitation in Reducing Early Neonatal Mortality and Morbidity
Brief Title: Neonatal Resuscitation With Supraglottic Airway Trial
Acronym: NeoSupra
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Centre For International Health (Other)
Collaborators: Makerere University (Other); University of Padova (Other); Karolinska Institutet (Other); Doctors with Africa - CUAMM (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NeoSupra
Record Dates: First submitted 2017-04-26; First posted 2017-04-28 (Actual); Last update posted 2020-06-29 (Actual); Status verified 2020-06

CONDITIONS: Asphyxia Neonatorum
MeSH Terms: conditions — Asphyxia Neonatorum | interventions — Masks

STUDY DESIGN:
Intervention Model Description: Day by day, infants will be randomized to either of the arms.
Who Masked: Outcomes Assessor
Masking Description: The neonatologists assessing the Thompson score will be blinded to the intervention arm. Other staff members will know about the arm allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Supraglottic airway (Experimental): All newborns in need of resuscitation in this arm will receive initial treatment with positive pressure ventilation using a supraglottic airway and a bag.
  Interventions: Device: Supraglottic airway
- Face-mask (Active Comparator): All newborns in need of resuscitation in this arm will receive initial treatment with positive pressure ventilation using a face-mask and a bag.
  Interventions: Device: Face-mask

INTERVENTIONS:
Device: Supraglottic airway — Instead of using a conventional face mask to provide positive pressure ventilation during neonatal resuscitation we are using a supraglottic airway and a conventional bag.
  Other Names: i-gel; supraglottic airway device
  Arms: Supraglottic airway
Device: Face-mask — In order to provide positive pressure ventilation during neonatal resuscitation we are using a conventional face-mask and a conventional bag.
  Arms: Face-mask

SUMMARY:
Mortality rates from birth asphyxia in low-income countries remain very high. Face mask ventilation (FMV) is the most common method of resuscitating neonates in such settings. It is mostly performed by midwives but may not always be satisfactory. The i-gel® is a cuffless supraglottic airway which is easy to insert and provides an efficient seal that prevents air leakage with the potential to enhance the performance of neonatal resuscitation. Midwives can be trained in a short time to use this method. A pilot study in Uganda has demonstrated that midwives can safely perform resuscitation of newborn with the i-gel.

OBJECTIVE To investigate whether the use of a cuffless supraglottic airway compared to face-mask ventilation during neonatal resuscitation can reduce early neonatal death (before 7 days of life) or morbidity in neonatal encephalopathy (NE) in asphyxiated neonates.

STUDY DESIGN, SETTING AND POPULATION A single-centre randomized clinical trial will be conducted at Mulago National Referral Hospital, Kampala, Uganda, among asphyxiated neonates in the delivery units. Prior to the intervention, all staff in the labour ward performing resuscitation will receive training according to the HBB curriculum with a special module for training on supraglottic airway insertion. Resuscitation will be performed according to international guidelines.

UTILITY OF THE STUDY It is crucial to explore alternative, cost-effective modalities that not only would reduce mortality, but also the burden of neurological damage in survivors.

DETAILED DESCRIPTION:
One of the targets in the SDG-3 is to reduce neonatal mortality to less than 12 per 1000 live births by 2030. This will require considerable effort in many low-income countries. Perinatal mortality contributes to 40% of infant mortality in Uganda. Early neonatal death from birth asphyxia (BA) could be as high 60%. New evidence-based strategies are needed to reduce mortality from BA in order to achieve SDG-3 by 2030.

Optimal care of the depressed newborn is crucial to prevent and manage BA. The challenge in low-income settings is that highly qualified staff is not readily available to attend to the newborn who require their expertise. In most cases, the midwives are the most skilled personal attending to deliveries and also responsible for resuscitating newborns. At present in low-income settings, FMV is the commonly used method for resuscitating depressed newborn. Easy-to-use equipment such as a supraglottic airway could contribute to obtain more effective ventilation, and improve the outcome of the infant.

This trial is based on a previous pilot trial ClinicalTrials.gov Identifier: NCT02042118.

Primary objective

• To assess if the proportion of either early neonatal death or neonatal encephalopathy (admission to NICU with a Thompson score of 11 or above in day 1-5 during hospitalisation), can be decreased from 40 % in the control arm (using FM) to 30 % or less in the intervention arm (using i-gel supraglottic airway), a 25% decrease.

Secondary objectives

* To assess the safety of a supraglottic airway in the hands of lower cadre (non-doctor) birth attendants in Africa.
* To assess if the proportion of very early and early neonatal deaths is lower in the intervention arm compared to the control arm.
* To assess if the proportion of neonatal encephalopathy (admission to NICU with maximum Thompson score 11 or above), is lower in the intervention arm compared to the control arm.
* To assess if the proportion of neonatal encephalopathy (admission to Neonatal Intensive Care Unit - NICU - with maximum Thompson score 7 or above), is lower in the intervention arm compared to the control arm.
* To assess if hospital admission rate in the first 7 days of life is lower in the intervention arm compared to the control arm.
* To assess the need of advanced resuscitation in the intervention arm compared to the control arm.

Study justification and significance

Training midwives and other birth-attendants can save lives. However, delivering effective positive pressure ventilation (PPV) with FM is a delicate task that requires continuous (re)training. In a previous phase II trial (NCT02042118), it has been shown that a supraglottic airway is safe to use, even in the hands of midwives and with the potential to deliver efficient PPV and perhaps even improve outcome of asphyxiated babies. The cuffless i-gel is simple to use and could therefore be the ideal device to resuscitate newborn when experienced physicians are not available.

Prior to interventions: training midwives in neonatal resuscitation skills

Helping Babies Breathe (HBB) is an evidence-based educational program to teach neonatal resuscitation techniques in resource-limited areas. It is an initiative of the American Academy of Pediatrics (AAP) in collaboration with the World Health Organization (WHO), US Agency for International Development (USAID), Saving Newborn Lives, the National Institute of Child Health and Development, and a number of other global health organizations.

The objective of HBB is to train birth attendants in developing countries in the essential skills of newborn resuscitation, with the goal of having at least one person who is skilled in neonatal resuscitation at the birth of every baby.

The second edition of HBB is now available and will be used in the training.

Study procedures

It is estimated that around 5-10 % of babies born will need ventilation as part of the resuscitation. This randomized trial will include all babies eligible for resuscitation. All newborns in need of resuscitation will be randomized to receive initial treatment using either:

* Supraglottic airway (intervention arm) or
* Face mask (active comparator arm).

The midwife will immediately move the babies not responding to stimulation to the resuscitation area. Ventilation with supraglottic airway or face mask will be initiated immediately. Apgar score and admission to the neonatal ward will be recorded by a research assistant. The intervention may be recorded on video to ensure quality assurance and data collection.

If the infant is hospitalised, daily assessment of Thompson score will be made by a skilled paediatrician/physician. A follow-up visit on day 7 (or later) will determine the outcome (if the infant is alive or not) together with the assessments of Thompson score.

ELIGIBILITY:
Inclusion Criteria:

* Inborn baby (=born in the hospital)
* Expected ≥ 34-week gestation
* Expected birth weight ≥ 2000 g
* Need for PPV at birth
* Parental consent

Exclusion Criteria:

* Major malformations (incompatible with sustained life or affecting the airways)

Max Age: 10 Minutes | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1163 (Actual)
Dates: Start 2018-05-08 (Actual); Primary Completion 2019-08-12 (Actual); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Composite outcome of either a) early neonatal death or b) neonatal encephalopathy | Day 7 of life
  A composite outcome of a) early neonatal death (within 7 days) b) neonatal encephalopathy (admission to NICU with a Thompson score of 11 or above in day 1-5 during hospitalisation).

SECONDARY OUTCOMES:
Number of adverse events (AEs) and serious adverse events (SAEs) | Day 7 of life
  Safety of i-gel in the hands of non-doctor birth attendants (AEs and SAEs)
Early neonatal death | Day 7 of life
  Early neonatal death (within 7 days)
Very early neonatal death | Day 1 of life
  Very early neonatal death (within 24 hours)
Neonatal encephalopathy | Day 7 of life
  Neonatal encephalopathy (admission to NICU with a Thompson score of 11 or above in day 1-5 during hospitalisation).
Mild neonatal encephalopathy | Day 7 of life
  Neonatal encephalopathy (admission to NICU with a Thompson score of 7 or above in day 1-5 during hospitalisation).
Any hospital admission | Day 7 of life
  Any hospital admission
Advanced resuscitation | Day 7 of life
  Advanced resuscitation including intervention by supervising physician

CONTACTS AND LOCATIONS:
Overall Officials: Thorkild Tylleskär, MD, PhD, Principal Investigator — University of Bergen, Norway
Locations (1):
- Mulago National Referral Hospital, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pejovic NJ, Trevisanuto D, Nankunda J, Tylleskar T. Pilot manikin study showed that a supraglottic airway device improved simulated neonatal ventilation in a low-resource setting. Acta Paediatr. 2016 Dec;105(12):1440-1443. doi: 10.1111/apa.13565. PMID 27582031
- [Background] Pejovic NJ, Trevisanuto D, Lubulwa C, Myrnerts Hook S, Cavallin F, Byamugisha J, Nankunda J, Tylleskar T. Neonatal resuscitation using a laryngeal mask airway: a randomised trial in Uganda. Arch Dis Child. 2018 Mar;103(3):255-260. doi: 10.1136/archdischild-2017-312934. Epub 2017 Sep 14. PMID 28912163
- [Background] Pejovic NJ, Myrnerts Hook S, Byamugisha J, Alfven T, Lubulwa C, Cavallin F, Nankunda J, Ersdal H, Segafredo G, Blennow M, Trevisanuto D, Tylleskar T. Neonatal resuscitation using a supraglottic airway device for improved mortality and morbidity outcomes in a low-income country: study protocol for a randomized trial. Trials. 2019 Jul 19;20(1):444. doi: 10.1186/s13063-019-3455-8. PMID 31324213
- [Derived] Larsson M, Myrnerts Hook S, Mpamize A, Tylleskar T, Lubulwa C, Trevisanuto D, Elfving K, Pejovic NJ. Oxygen saturation after birth in resuscitated neonates in Uganda: a video-based observational study. BMJ Paediatr Open. 2022 Jan;6(1):e001225. doi: 10.1136/bmjpo-2021-001225. PMID 35258476
- [Derived] Pejovic NJ, Myrnerts Hook S, Byamugisha J, Alfven T, Lubulwa C, Cavallin F, Nankunda J, Ersdal H, Blennow M, Trevisanuto D, Tylleskar T. A Randomized Trial of Laryngeal Mask Airway in Neonatal Resuscitation. N Engl J Med. 2020 Nov 26;383(22):2138-2147. doi: 10.1056/NEJMoa2005333. PMID 33252870